CLINICAL TRIAL: NCT00853125
Title: Phase II Study of Sunitinib Plus Extended Courses of Irradiated Allogeneic Lymphocytes for Patients With Renal Cell Carcinoma (SPECIAL Trial)
Brief Title: Sunitinib and Irradiated Donor Lymphocytes in Treating Patients With Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Roger Strair, MD, PhD, Professor of Medicine, RWJMS, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0220080220; P30CA072720 (NIH); CDR0000635763 (Other: NCI); 0220080220 (Other: IRB); 080708 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib plus Irradiated Allogeneic Lymphocytes (Experimental)
  Interventions: Biological: therapeutic allogeneic lymphocytes; Drug: sunitinib malate

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes — Patients with a partially HLA-matched family member who can serve as a hematopoietic stem cell transplant donor will receive partially HLA-matched irradiated donor lymphocytes approximately every 8 weeks depending upon response
Drug: sunitinib malate — Sunitinib will be administered orally at a dose of 50 mg qd for 4 consecutive weeks followed by 2 weeks off for every cycle.

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Infusing irradiated donor lymphocytes into the patient may help the patient's immune system kill tumor cells. Giving sunitinib together with irradiated donor lymphocytes may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving sunitinib together with irradiated donor lymphocytes works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine progression-free survival of patients with metastatic clear cell renal cell carcinoma treated with sunitinib and irradiated allogeneic lymphocytes.

Secondary

* Determine rates and kinetics of clinical/radiographic response in these patients.
* Determine toxicities associated with treatment in these patients.
* Assess stable disease at 6 months in these patients.
* Assess overall survival of these patients.

OUTLINE: Patients receive oral sunitinib malate once daily for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Beginning with course 2 of sunitinib malate, patients also receive irradiated allogeneic lymphocytes IV over 1 hour every 8-16 weeks for up to 6 infusions in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 60 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Primary lesion or metastatic site demonstrating clear cell variant with < 25% of any other histology
* Radiographically measurable disease by RECIST criteria
* Initiated treatment with sunitinib malate ≤ 6 weeks ago
* No radiographically detectable brain metastases by MRI or CT scan
* HLA-partially matched related donor available, as determined by serologic and/or DNA typing

  * Appropriate HLA match (≥ 2/6 HLA A, B, DR match)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Total bilirubin ≤ 2.0 times upper limit of normal (ULN)
* AST ≤ 3.0 times ULN
* Calculated creatinine clearance ≥ 40 mL/min
* Cardiac ejection fraction ≥ 50%
* QTc interval < 500 msec by EKG
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* None of the following within the past 6 months:

  * Myocardial infarction
  * Severe/unstable angina
  * Coronary/peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
* No ongoing ventricular cardiac dysrhythmias ≥ grade 2, according to NCI CTCAE v3.0
* No history of serious ventricular arrhythmia (e.g., ventricular tachycardia > 3 beats in a row)
* No ongoing atrial fibrillation
* No other malignancies within the past 3 years, other than basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, or ductal or lobular carcinoma in situ of the breast
* No other concurrent serious illness

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic therapy for metastatic renal cell carcinoma
* No prior immunotherapy
* No prior VEGF-targeted or mTOR-targeted therapies
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital), St. John's wort, ketoconazole, dexamethasone, dysrhythmic drugs (e.g., terfenadine, quinidine, procainamide, sotalol, probucol, bepridil, indapamide, or flecainide), haloperidol, risperidone, rifampin, grapefruit, or grapefruit juice
* No other concurrent investigational anticancer agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2014-02-22 (Actual); Study Completion 2014-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey. The study was open to accrual on 02/03/2009 and closed to accrual on 05/07/2013 because of slow accrual.
Pre-assignment Details: We are reporting results on 10 eligible patients. Five patients were deemed ineligible.
Period: Overall Study
Arm/Group | Sunitinib Plus Irradiated Allogeneic Lymphocytes
Started | 10
Completed | 9
Not Completed | 1
Not completed — Study participant's donor was CMV + | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib Plus Irradiated Allogeneic Lymphocytes
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Determined as the time from treatment with combination sunitinib with irradiated allogeneic lymphocytes to progressive disease or death whichever occurred first. Progression is determined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v 1.0) as 20% increase in the sum of the of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, on average up to 1 year.
Population: Study was terminated early due to slow accrual.
Measure: Median (Full Range); unit: days
Arm/Group | Sunitinib Plus Irradiated Allogeneic Lymphocytes
Number analyzed (Participants) | 7
days | 137 [15 to 489]

2. Secondary Outcome: Response Rate
Description: Per response evaluation criteria in solid tumors criteria (RECIST v 1.0) for target lesions and assessed by MRI; Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; Stable disease - not meeting criteria for response or progression.
Time Frame: Best responseFrom date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year.
Measure: Number; unit: participants
Groups:
- Sunitinib Plus Irradiated Allogeneic Lymphocytes: Therapeutic Allogeneic Lymphocytes: patients with a partially HLA-matched family member who can serve as a hematopoietic stem cell transplant donor will receive partially HLA-matched irradiated donor lymphocytes approximately every 8 weeks depending upon response.
  Sunitinib malate: Sunitinib will be administered orally at adose 50 mg qd for 4 consecutive weeks followed by 2 weeks off for every cycle.
Arm/Group | Sunitinib Plus Irradiated Allogeneic Lymphocytes
Number analyzed (Participants) | 10
participants
  PR | 3
  Progressive Disease | 2
  Stable Disease | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 336 days per patient.
Arm/Group | Sunitinib Plus Irradiated Allogeneic Lymphocytes
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes